CLINICAL TRIAL: NCT05562297
Title: A Phase II Study to Evaluate the Safety and Efficacy of Sintilimab Combined With Nab-paclitaxel and Gemcitabine for Neoadjuvant and Adjuvant Therapy of Patients With Resectable and Borderline Resectable Pancreatic Cancer
Brief Title: Neoadjuvant/Adjuvant Sintilimab, Nab-paclitaxel, and Gemcitabine for Resectable/Borderline Resectable Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSPAC-01
Record Dates: First submitted 2022-09-20; First posted 2022-09-30 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer, Stage IB; Pancreatic Cancer, Stage IIA; Pancreatic Cancer, Stage IIB; Pancreatic Cancer Stage III
Keywords: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; Sintilimab; Nab-paclitaxel; Gemcitabine; Neoadjuvant Therapy; Adjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — sintilimab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sintilimab + nab-paclitaxel + gemcitabine (Experimental): Experimental: sintilimab + nab-paclitaxel + gemcitabine nab-paclitaxel at 125 mg/m^2 on days 1, and 8; gemcitabine at 1000 mg/m^2 on days 1, and 8; sintilimab at 200mg on day 1;
  Interventions: Drug: sintilimab; Drug: nab-paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: sintilimab — Patients firstly receive sintilimab 200 mg (iv, 30 minutes) on day 1 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 3 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: Tyvyt
Drug: nab-paclitaxel — Patients firstly receive nab-paclitaxel 125 mg/m^2 (iv, 30 minutes) on days 1, and 8 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 3 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: Abraxane
Drug: gemcitabine — Patients secondly receive gemcitabine 1000 mg/m^2 (iv, 30 minutes) on days 1, and 8 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 3 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: GEMZAR

SUMMARY:
The purpose of this research is to investigate the activity and safety of the combination of gemcitabine plus nab-paclitaxel and sintilimab as neoadjuvant therapy in treating patients with resectable and borderline resectable pancreatic cancer.

The drugs involved in this study are:

* Sintilimab
* Nab-paclitaxel
* Gemcitabine

DETAILED DESCRIPTION:
Pancreatic cancer is a highly fatal disease with a 5-year survival rate of less than 5%, and it is becoming an increasingly common cause of cancer mortality. Neoadjuvant therapy, such as gemcitabine plus nab-paclitaxel, can effectively avoid the proliferation of residual tumors and reduce the risk of lymph node metastasis, implantation metastasis during surgery, and early relapse after operation. Most importantly, it can change the immune status by turning the "immune cold" pancreatic cancer into an "immune hot" condition, which will enable the application of immune checkpoint inhibitors. Sintilimab is an immune checkpoint inhibitor against programmed cell death protein 1, which is applicable for treatment of a range of cancers including non-small cell lung cancer, melanoma, esophageal cancer, and liver cancer. It could block the interaction between PD-1 and its ligands and help the anti-tumor effect of T cells to recover. The present study is intended to investigate the activity and safety of the combination of gemcitabine plus nab-paclitaxel and sintilimab as neoadjuvant therapy in treating patients with resectable and borderline resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥ 18 years and ≤ 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have imaging evaluations to confirm that their pancreatic adenocarcinoma is resectable and borderline resectable. Patients must have histologically confirmed pancreatic adenocarcinoma, too.
* Therapy-naïve for their pancreatic cancer. Patients should receive no anti-tumor treatment, including systemic chemotherapy, interventional chemotherapy, high-energy focused ultrasound, radiotherapy, immunotherapy, molecular targeted therapy, and anti-tumor Chinese medicine therapy.
* No serious dysfunction in blood system, heart, lung function, or autoimmune system (refer to the respective diagnostic criteria)
* White blood cell (WBC) ≥ 3 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets (PLT) ≥ 100 × 109/L; Hemoglobin (Hgb) ≥ 90 g/L
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 × institutional upper limit of normal (ULN); Total bilirubin (TBIL) ≤ ULN; Creatinine (CRE) ≤ 1.5 × ULN
* Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 × ULN
* Able to comply with research visit plans and other protocol requirements.

Exclusion Criteria:

* The diameter of the resectable tumor is ≤ 2 cm in imaging evaluation
* Associated with other malignant tumors
* Patients receiving anti-tumor treatment before neoadjuvant therapy, including systemic chemotherapy, interventional chemotherapy, high-energy focused ultrasound, radiotherapy, immunotherapy, molecular targeted therapy, and anti-tumor Chinese medicine therapy
* Use of any other investigational agents
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, internal hemorrhage, pancreatic leakage, bile leakage, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing women
* History of allergic reactions attributed to compounds of similar chemical or biological composition to nab-paclitaxel, gemcitabine, or sintilimab
* Patients who are using and need to use warfarin for a long period
* Patients who are unwilling or unable to comply with study procedures
* Patients who are expected to be out of the observation period for 14 days or more during the treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival after the application of sintilimab and gemcitabine plus nab-paclitaxel | From date of enrollment to the date of death for any cause, assessed 2 months during therapy and 3 months thereafter up to 24 months
  To evaluate the overall survival of patients with resectable and borderline resectable pancreatic cancer treated with the combination of sintilimab and gemcitabine plus nab-paclitaxel. Outpatient visit, phone interview

SECONDARY OUTCOMES:
Overall survival after the application of sintilimab and gemcitabine plus nab-paclitaxel | From date of enrollment until the date of death from any cause, assessed one month during therapy and 3 months thereafter up to 24 months
  To evaluate the overall survival of patients treated with this regimen. Outpatient visit, phone interview
Event-free survival after the application of sintilimab and gemcitabine plus nab-paclitaxel | From date of enrollment until the date of death from any cause, assessed one month during therapy and 3 months thereafter up to 24 months
  To evaluate the event-free survival of patients treated with this regimen. Outpatient visit, phone interview
Objective response rate and disease control rate after finishing the course of the treatment of sintilimab and gemcitabine plus nab-paclitaxel | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the objective response rate and disease control rate of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Recurrence-free survival after finishing the course of the treatment of sintilimab and gemcitabine plus nab-paclitaxel and curative resection | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the recurrence-free survival of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Resection rate and R0 resection rate after finishing the course of the treatment of sintilimab and gemcitabine plus nab-paclitaxel and curative resection | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the resection rate and R0 resection rate of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Major pathological response rate after finishing the course of the treatment of sintilimab and gemcitabine plus nab-paclitaxel and curative resection | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the major pathologic response rate of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Node-negative resection rate, the occurrence rate and severity of perioperative complications after finishing the course of the treatment of sintilimab and gemcitabine plus nab-paclitaxel and curative resection | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the node-negative resection rate, the occurrence rate and severity of perioperative complications of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Progression-free survival after finishing the course of the treatment of sintilimab and gemcitabine plus nab-paclitaxel, but being determined as unresectable after surgical exploration | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the progression-free survival of patients treated with this regimen, but determined as unresectable after surgical exploration. Outpatient visit, phone interview
Number and severity of toxicities according to NCI CTCAE version 4.0 | One week during therapy and 3 months thereafter up to 24 months
  To evaluate the occurrence of toxicities according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE; version 4.0) in patients treated with this regimen. The toxicity profile includes but not limits neutropenia, thrombocytopenia, peripheral neuropathy, hypoglycemia, metabolic acidosis (acute or chronic, including ketoacidosis), which will be summarized as the percentage of patients by type and grade according to treatment group. Outpatient visit, phone interview, laboratory findings
Correlation between patients' immunological parameters before and after the application of sintilimab and gemcitabine plus nab-paclitaxel and prognosis of them | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the correlation between status of immunological parameters (such as MSI, TMB, the expression of PD-1/PD-L1, and dMMR) and prognosis of patients treated with this regimen. Outpatient visit, laboratory findings
Whole exome sequencing before and after the application of sintilimab and gemcitabine plus nab-paclitaxel | One month before therapy and one month after therapy
  To evaluate difference of the whole exome sequencing before and after the therapy. To evaluate the relation between the difference of whole exome sequencing and immunological parameters of patients treated with this regimen. To evaluate the relation between the difference of whole exome sequencing and the prognosis of patients treated with this regimen. Outpatient visit, laboratory findings
Correlation between circulating tumor DNA (ctDNA) and serum tumor marker before and after neoadjuvant therapy, before and after curative resection, during and after adjuvant therapy, and during and after the maintenance treatment of immunotherapy | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the correlation between ctDNA and serum tumor markers, such as CA199, CA125, and CEA levels of patients. Outpatient visit, laboratory findings
Correlation between ctDNA and CT evaluations before and after neoadjuvant therapy, before and after curative resection, during and after adjuvant therapy, and during and after the maintenance treatment of immunotherapy | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the consistency between ctDNA and CT evaluations of patients. Outpatient visit, laboratory findings
Correlation among ctDNA, serum tumor markers, and CT evaluations before and after neoadjuvant therapy, before and after curative resection, during and after adjuvant therapy, and during and after the maintenance treatment of immunotherapy. | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the correlation among ctDNA, serum tumor markers, and CT evaluations of patients. Outpatient visit, laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Liang Liu, MD, PhD, Principal Investigator — Shanghai Zhongshan Hospital; Wen-hui Lou, MD, PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers in order to protect patients' privacy.